CLINICAL TRIAL: NCT07239973
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single/Multiple-dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BGM0504 Tablets Orally Administered in Healthy and Non-diabetic Overweight or Obese Chinese Subjects.
Brief Title: A Study of BGM0504 Tablets in Healthy and Non-diabetic Overweight or Obese Chinese Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-CPK-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Non-diabetic Overweight or Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGM0504 tablets (Experimental): Oral administration once daily
  Interventions: Drug: BGM0504 tablets
- Placebo tablets (Experimental): Placebo Oral administration once daily
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: BGM0504 tablets — Administered p.o.
  Arms: BGM0504 tablets
Drug: Placebo tablets — Administered p.o.
  Arms: Placebo tablets

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Single/Multiple-dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BGM0504 Tablets Orally Administered in Healthy and Non-diabetic Overweight or Obese Chinese Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years (inclusive) at the time of screening , healthy and non-diabetic overweight or obese subjects , both male and female;
* Healthy subjects , male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 20.0 kg/m² ≤ BMI < 28 kg/m²（BMI = weight/height²）;
* Obese individuals: BMI ≥ 28.0 kg/m², or overweight individuals: 24.0 kg/m² ≤ BMI < 28.0 kg/m²;
* (Medical Inquiry) Have a stable body weight (<5% self-reported change during the previous 12 weeks) before screening.
* Have no history of mental disorders, be able to communicate smoothly with Investigator, Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.
* Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subject) plus an additional medically acceptable form of contraception (female partner) for the duration of the study and for at least 3 months after dosing; must also agree to refrain from sperm donation for at least 3 months post dose

Exclusion Criteria:

* Those with a history of severe drug allergies (especially those with known or suspected allergies to the active ingredients and excipients of BGM0504 Tablets), or complicated with severe specific allergic diseases/history, or with a severe allergic constitution.
* Subjects with positive results for HBsAg, anti-HCV, anti-HIV or anti-TP during the screening period.
* At the screening/baseline period, any one of the laboratory test indicators meets the following criteria:

  1. fasting serum glucose≥ 7.0mmol/L, or post-prandial glucose (PPG)-2h≥ 11.1mmol/L in oral glucose tolerance test (OGTT); (During screening, participants with fasting serum glucose ranging from 6.1 to 6.9mmol/L shall undergo the OGTT.)
  2. ALT, AST ≥ 2.5 times upper limit of normal (ULN) or total bilirubin ≥ 1.5 times upper limit of normal (ULN)
  3. Glomerular filtration rate (eGFR) ≤ 80 mL/min/1.73 m2(using CKD-EPI formula) or positive urine protein 2+ or more.
  4. Serum calcitonin level ≥ 35 ng/L (pg/mL);
  5. Thyroid-stimulating hormone (TSH) > 6.0mIU/L or < 0.4mIU/L;
  6. Fasting triglycerides ≥ 5.64mmol/L (500 mg/dL);
  7. Hemoglobin (Hgb) < 100 g/L (for females) or < 110 g/L (for males);
* 12-lead ECG shows ventricular heart rate < 50 beats/min or > 100 beats/min at screening/baseline, second or third degree atrioventricular block, long QT syndrome, QTcF> 470ms for women or > 450ms for men, pre-excitation syndrome or other significant arrhythmias.
* Used illegal drugs within 6 months prior to screening, or substance abuse within 12 months prior to screening.
* Participated in drug or medical device clinical trials and treated with Study Drug (excluding placebo) or medical device intervention within 12 weeks before screening.
* Participants who have received any vaccine within 2 weeks prior to screening, or plan to receive a vaccine during the trial.
* Female participants who are pregnant or lactating, or those with a positive pregnancy test result during the screening period.
* Positive urine drug test or alcohol serum test result at screening or at baseline.
* Has any other conditions or disorders deemed unsuitable for including in the study, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of treatment adverse events | 8 weeks
  The relationship of each adverse event to the investigational product was assessed by the investigator

SECONDARY OUTCOMES:
Pharmacokinetic endpoint: Concentration of BGM0504 in plasma | 8 weeks
Change in fasting weight at week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Yunnan University of Chinese Medicine, Kunming, Yunnan, China